CLINICAL TRIAL: NCT03053102
Title: A Phase 2 Open-Label Proof of Concept Study to Assess the Efficacy, Safety, and Pharmacokinetics of ACH-0144471 in Untreated Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Study of Danicopan in Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH471-100; 2016-002652-25 (EudraCT Number); U1111-1190-3490 (Other: UTN)
Record Dates: First submitted 2017-02-01; First posted 2017-02-14 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: PNH; Paroxysmal; Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemoglobinuria | interventions — danicopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Danicopan (Experimental): Starting doses of danicopan ranged from 100 to 150 milligrams (mg) three times daily (TID), with subsequent dose escalation up to 200 mg TID based on response (clinical and biochemical) for 28 days (Part 1). Participants with reductions in lactate dehydrogenase (LDH) meeting specified criteria were offered continued dosing beyond Day 28, for up to 8 additional weeks (Part 2).
  Interventions: Drug: Danicopan

INTERVENTIONS:
Drug: Danicopan — Danicopan was administered as multiple oral doses over a period of at least 28 days.
  Other Names: ACH-0144471; ACH-4471; ACH4471; 4471; ALXN2040

SUMMARY:
The purpose of this study was to determine the safety and efficacy of ACH-0144471 (also known as danicopan and ALXN2040) in currently untreated participants with PNH.

DETAILED DESCRIPTION:
After 12 weeks of treatment, participants deriving clinical benefit were offered enrollment in a separate long-term extension study (ACH471-103, NCT03181633).

ELIGIBILITY:
Inclusion Criteria:

* Currently untreated PNH participants with PNH Type III erythrocyte and/or granulocyte clone size ≥10% and anemia (hemoglobin <12 grams/deciliter) with adequate reticulocytosis (as determined by the Investigator).
* LDH ≥1.5 x the upper limit of normal.
* Platelets ≥50,000/microliter without the need for platelet transfusions.
* Documentation of vaccination for Neisseria meningitidis, Haemophilus influenza, and Streptococcus pneumoniae, or willingness to receive vaccinations during the screening period.
* Negative pregnancy test for females prior to dosing and throughout the study.

Exclusion Criteria:

* History of a major organ transplant (for example, heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Participants who had received another investigational agent within 30 days or 5 half-lives of the investigational agent prior to study entry, whichever is greater.
* Participants who had received eculizumab at any dose or interval within the past 75 days before study entry.
* Participants with known or suspected complement deficiency.
* Participants with active bacterial infection or clinically significant active viral infection, a body temperature >38°Celsius, or other evidence of infection on Day 1, or with a history of febrile illness within 14 days prior to first study drug administration.
* History of meningococcal infection, or a first-degree relative or household contact with a history of meningococcal infection.
* Females who were pregnant, nursing, or planning to become pregnant during the study or within 90 days of study drug administration or participants with a female partner who was pregnant, nursing, or planning to become pregnant during the study or within 90 days of study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (2):
  - Clinical Trial Site, Florence
  - Clinical Trial Site, Naples
- Clinical Trial Site, Auckland, New Zealand
- Clinical Trial Site, Seoul, South Korea
- Clinical Trial Site, London, United Kingdom

REFERENCES:
- [Result] Risitano AM, Kulasekararaj AG, Lee JW, Maciejewski JP, Notaro R, Brodsky R, Huang M, Geffner M, Browett P. Danicopan: an oral complement factor D inhibitor for paroxysmal nocturnal hemoglobinuria. Haematologica. 2021 Dec 1;106(12):3188-3197. doi: 10.3324/haematol.2020.261826. PMID 33121236

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 2 parts. In Part 1, participants received danicopan for 28 days. Starting doses were 100 or 150 milligrams (mg) three times daily (TID). A further dose increase up to 175 mg TID (N=8 participants) and 200 mg TID (N=4 participants) was conducted. Participants with reductions in lactate dehydrogenase (LDH) meeting specified criteria were offered continued dosing beyond Day 28, for up to 8 additional weeks (Part 2).
Groups:
- Danicopan: Participants received danicopan 100 to 200 mg TID.
Period: Study Part 1: 28-Day Treatment
Arm/Group | Danicopan
Started | 10
Received at Least 1 Dose of Study Drug | 10
Completed | 10
Not Completed | 0
Period: Study Part 2: 84-Day Treatment
Arm/Group | Danicopan
Started | 10
Completed | 8
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study and received at least 1 dose of study drug.
Arm/Group | Danicopan
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.94 (13.575)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Other | 1
Region of Enrollment [Number; unit: participants]
  New Zealand | 6
  South Korea | 1
  United Kingdom | 1
  Italy | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Serum LDH Levels At Day 28
Description: Change from Baseline = Serum LDH levels on Day 28 - Baseline Serum LDH levels.
Time Frame: Baseline, Day 28
Population: All participants who received at least 1 dose of study drug and had analyzable data at the timepoints specified.
Measure: Mean (Standard Deviation); unit: international units per liter (IU/L)
Arm/Group | Danicopan
Number analyzed (Participants) | 10
international units per liter (IU/L)
  Baseline | 1416 (540.25)
  Day 28 (Part 1) | 444.3 (255.78)
  Change from Baseline | -971.7 (549.76)

2. Secondary Outcome: Change From Baseline In Hemoglobin (Hgb) At Days 28 And 84
Description: Change from Baseline = Hgb levels on Days 28 or 84 - Baseline Hgb levels.
Time Frame: Baseline, Days 28 and 84
Population: All participants who received at least 1 dose of study drug and had analyzable data at the timepoints specified.
Measure: Mean (Standard Deviation); unit: grams/deciliter (g/dL)
Arm/Group | Danicopan
Number analyzed (Participants) | 10
grams/deciliter (g/dL)
  Baseline | 9.76 (1.758)
  Part 1: Day 28 | 10.94 (1.651)
  Part 1: Change from Baseline at Day 28 | 1.18 (0.877)
  Part 2: Day 84: number analyzed (Participants) | 8
  Part 2: Day 84 | 11.45 (1.414)
  Part 2: Change from Baseline at Day 84: number analyzed (Participants) | 8
  Part 2: Change from Baseline at Day 84 | 1.80 (1.166)

3. Secondary Outcome: Change From Baseline In Serum LDH Levels At Day 84
Description: Change from Baseline = Serum LDH levels on Day 84 - Baseline Serum LDH levels.
Time Frame: Baseline, Day 84
Population: All participants who received at least 1 dose of study drug and had analyzable data at the timepoints specified.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Danicopan
Number analyzed (Participants) | 10
IU/L
  Baseline | 1416 (540.25)
  Day 84 (Part 2): number analyzed (Participants) | 8
  Day 84 (Part 2) | 537.3 (260.42)
  Change from Baseline: number analyzed (Participants) | 8
  Change from Baseline | -865.9 (447.86)

4. Secondary Outcome: Paroxysmal Nocturnal Hemoglobinuria (PNH) Type III Red Blood Cell (RBC) Clone Size
Description: PNH RBC, summed type III, clone size levels were assessed from Baseline to Day 28 and Day 84. The PNH clone size refers to the percentage of PNH-affected cells versus normal cells within the total cell population.
Time Frame: Baseline, Day 28, and Day 84
Population: All participants who received at least 1 dose of study drug and had analyzable data at the timepoints specified.
Measure: Mean (Standard Deviation); unit: percentage of the total cell population
Arm/Group | Danicopan
Number analyzed (Participants) | 10
percentage of the total cell population
  Baseline | 31.5363 (24.62004)
  Day 28: number analyzed (Participants) | 9
  Day 28 | 43.6279 (15.58021)
  Day 84: number analyzed (Participants) | 8
  Day 84 | 56.2953 (19.85086)

5. Secondary Outcome: Serious Adverse Events (SAEs), Grade 3 And Grade 4 Treatment-emergent Adverse Events (TEAEs), And Adverse Events (AEs) Leading To Discontinuation
Description: An AE was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), important medical event or reaction. The intensity of an AE was graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Adverse Event Severity Grading Table. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: After the first dose of study medication (Day 1) through 14 days after the last dose of study drug (up to Day 104)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Danicopan
Number analyzed (Participants) | 10
Participants
  SAE | 1
  TEAE Grade 3 | 1
  TEAE Grade 4 | 1
  AE leading to discontinuation | 1

6. Secondary Outcome: Grade 3 And Grade 4 Laboratory Abnormalities
Description: Laboratory abnormalities were determined from laboratory measurements analyzed at the central or local laboratories, and were graded using CTCAE.
Time Frame: After the first dose of study medication (Day 1) through 14 days after the last dose of study drug (up to Day 104).
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Danicopan
Number analyzed (Participants) | 10
Participants
  Alanine aminotransferase increased | 1
  Aspartate aminotransferase increased | 1
  Low hemoglobin | 1
  Low neutrophil count | 4
  High triglycerides | 1

7. Secondary Outcome: Pharmacokinetics (PK): Area Under The Plasma Concentration-time Curve From Time Of Administration To 8 Hours Post-dose (AUC0-8)
Description: Serial blood samples were collected predose and up to 8 hours postdose.
Time Frame: Days 6 and 20
Population: All participants who received at least 1 dose of study drug and had analyzable data at the timepoints specified. PK analysis was not conducted on the 200 mg dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (hr)*nanograms/milliliter (ng/mL)
Arm/Group | Danicopan
Number analyzed (Participants) | 10
hour (hr)*nanograms/milliliter (ng/mL)
  Day 6: 100 mg TID: number analyzed (Participants) | 2
  Day 6: 100 mg TID | 1432.611 (19.41)
  Day 20: 150 mg TID: number analyzed (Participants) | 4
  Day 20: 150 mg TID | 2370.421 (14.92)
  Day 20: 175 mg TID: number analyzed (Participants) | 6
  Day 20: 175 mg TID | 2278.038 (37.30)

8. Secondary Outcome: PK: Maximum Plasma Concentration (Cmax)
Description: Serial blood samples were collected predose and up to 12 hours postdose.
Time Frame: Days 6 and 20
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Danicopan
Number analyzed (Participants) | 10
ng/mL
  Day 6: 100 mg TID: number analyzed (Participants) | 2
  Day 6: 100 mg TID | 347.707 (9.57)
  Day 20: 150 mg TID: number analyzed (Participants) | 4
  Day 20: 150 mg TID | 583.626 (27.29)
  Day 20: 175 mg TID: number analyzed (Participants) | 6
  Day 20: 175 mg TID | 516.8788 (33.39)

9. Secondary Outcome: PK: Time To Maximum Concentration (Tmax)
Description: Serial blood samples were collected predose and up to 12 hours postdose.
Time Frame: Days 6 and 20
Population: as for outcome 7
Measure: Median (Full Range); unit: hr
Groups:
- Danicopan: Participants who received danicopan 100 to 200 mg TID.
Arm/Group | Danicopan
Number analyzed (Participants) | 10
hr
  Day 6: 100 mg TID: number analyzed (Participants) | 2
  Day 6: 100 mg TID | 4.17 [3.67 to 4.67]
  Day 20: 150 mg TID: number analyzed (Participants) | 4
  Day 20: 150 mg TID | 3.67 [1.05 to 4.67]
  Day 20: 175 mg TID: number analyzed (Participants) | 6
  Day 20: 175 mg TID | 4.11 [1.67 to 4.65]

10. Secondary Outcome: Complement Alternative Pathway (AP) Functional Activity
Description: Serum AP functional activity was measured by the Wieslab functional immunoassay method.
Time Frame: Baseline and Day 28
Population: All participants who received at least 1 dose of study drug and had analyzable data at the timepoints specified.
Measure: Mean (Standard Deviation); unit: percentage of activity
Arm/Group | Danicopan
Number analyzed (Participants) | 10
percentage of activity
  Baseline | 65.216 (13.7143)
  Day 28 | 12.730 (14.37670)

11. Secondary Outcome: Complement Bb
Description: Plasma Bb was measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline and Day 28
Population: All participants who received at least 1 dose of study drug and had analyzable data at the timepoints specified.
Measure: Mean (Standard Deviation); unit: microgram (ug)/mL
Arm/Group | Danicopan
Number analyzed (Participants) | 10
microgram (ug)/mL
  Baseline | 2.24160 (0.773962)
  Day 28 | 0.83913 (0.838219)

ADVERSE EVENTS:
Time Frame: After the first dose of study medication (Day 1) through 14 days after the last dose of study drug (up to Day 104).
Description: [Not specified]
Arm/Group | Danicopan
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Danicopan (N=10)
Haemolysis (Blood and lymphatic system disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Danicopan (N=10)
Back pain (Musculoskeletal and connective tissue disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Headache (Nervous system disorders) | 4
Viral upper respiratory tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Fatigue (General disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Irritability (Psychiatric disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vaccination site erythema (General disorders) | 1
Paroxysmal nocturnal haemoglobinuria (Blood and lymphatic system disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1/5
Haemoglobinuria (Renal and urinary disorders) | 2
Haemolysis (Blood and lymphatic system disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pharyngitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT03053102/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT03053102/SAP_001.pdf